CLINICAL TRIAL: NCT02141022
Title: A Pilot Study of Plasticity-Based and Adaptive Cognitive Remediation in Adults With Multiple Sclerosis Treated With Gilenya
Brief Title: Computerized Exercise Training for Cognitive Remediation in Adults With Multiple Sclerosis Treated With Gilenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Lauren Krupp, Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DUS26T; IIRP-1450
Record Dates: First submitted 2014-02-14; First posted 2014-05-16 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Sclerosis; Cognitive Deficits; Gilenya Modifying Therapy for MS
Keywords: Multiple Sclerosis; Cognition; Cognitive Remediation; Gilenya; Computerized Cognitive Exercise
MeSH Terms: conditions — Multiple Sclerosis; Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PACR Program: Plasticity based, Adaptive Cognitve Remediation (Experimental): PACR Program Use: To use PACR, the participant navigates to the PACR study web site. The participant then logs into the PACR (using a study provided screen name and study identification number). A game-like experience begins, where the participant is presented with games in a set order. Each game consists of targeted exercises that contain the core science stimuli and tasks. The scheduling mechanism ensures that a participant progresses through the exercises in a defined order, generally moving from more simple (early sensory processing) exercises to more complex (multimodal, cognitive control) exercises over the course of the three-month experience.
  Interventions: Other: plasticity-based computerized cognitive remediation program; Drug: Gileyna
- Ordinary Computer Games (Active Comparator): Active Control Program Use (Ordinary Computer Games): The active control program is composed of 13 ordinary computer games matched to the PACR condition overall. This condition is designed to be a face-valid approach to cognitive remediation. The control condition is also designed to account for nonspecific treatment effects, including placebo response, interactions with research personnel, and experience with computers and computer-related activities, and any halo or expectation effect on study assessments.
  Interventions: Drug: Gileyna

INTERVENTIONS:
Other: plasticity-based computerized cognitive remediation program
  Arms: PACR Program: Plasticity based, Adaptive Cognitve Remediation
Drug: Gileyna

SUMMARY:
This study is investigating the efficacy of computer-based cognitive exercises as a means of cognitive remediation in patients with Multiple Sclerosis (MS) who are beginning the disease modifying pharmacotherapy Gileyna.

DETAILED DESCRIPTION:
Gilenya represents the most recent advance in MS disease-modification therapy (DMT) and shows promise for neuroprotection, a feature relevant to the progressive neurologic damage associated with the disease. Cognitive impairment accompanies MS in 40-60% of cases and when present, additional symptomatic treatment combined with DMT is required. To date no symptomatic pharmacologic therapy has shown a consistent benefit on MS associated cognitive dysfunction. However, non-pharmacologic approaches show promise. With recent technical and scientific advances, cognitive training is rapidly evolving to become the most effective intervention for the cognitive impairments associated with a wide range of neurological conditions. However, these training programs have not yet been studied in MS.

This study will be a randomized open-label clinical pilot trial to compare a plasticity-based and adaptive cognitive remediation (PACR) program to an active control (ordinary computer games) in 20 adults with multiple sclerosis (MS) starting Gilenya therapy. Primary outcome measures will be used as preliminary indicators of effect, with improvements on program task-related measures and changes in cognitive measures. Secondary outcome measures will determine the feasibility of the use of these programs in patients with MS, as indicated by compliance and patient-reported experience.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* Relapsing Remitting MS Diagnosis [81]
* Initiating Gilenya therapy, or current Gilenya therapy (kept constant for the past one month)
* No relapse or steroids in previous month
* Reading score on WRAT-3 of 37 or greater
* Visual, auditory and motor capacity to operate computer software, as judged by treating neurologist or study staff.

Exclusion Criteria:

* Previous trial of Gilenya therapy
* History of mental retardation, pervasive developmental disorder or other neurological condition associated with cognitive impairment
* Primary psychiatric disorder or unstable medical disorder that would influence ability to participate
* History of computer-based training with procedures similar to those proposed
* Learned English language after 12 years of age
* Unable to comply with study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Neuropsychological Test Results at 12weeks | 12 weeks

SECONDARY OUTCOMES:
Evaluate the feasibility of PACR for adults with MS on Gilenya therapy who have cognitive impairment based on Participant Adherence to Study Protocol | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Krupp, M.D., Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No